CLINICAL TRIAL: NCT06152588
Title: Restricted Eating Time in the Treatment of Type 2 Diabetes - the RESET2 Trial.
Brief Title: Restricted Eating Time in the Treatment of Type 2 Diabetes
Acronym: RESET2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University of Leeds (Other); Salk Institute for Biological Studies (Other); University of Copenhagen (Other); Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-23035125
Record Dates: First submitted 2023-10-27; First posted 2023-11-30 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
Keywords: Time-restricted eating; Type 2 Diabetes; Obesity; Overweight; Fasting; Circadian rhythm
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Fasting; Obesity; Overweight; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Time-restricted eating (Experimental): TRE group for 1 year: The intervention consists of a 3-month (12 weeks) strict TRE period, where participants follow the same eating window each day with minimal support, followed by a 9-month (40 weeks) period of individually adjusted TRE according to their experiences.
  Interventions: Other: Time restricted eating
- Control (No Intervention): Control group for 1 year: Participants will be instructed to continue their habitual lifestyle during the study and they will follow standard care with regular visits at the SDCC clinic 3-4 times/year.

INTERVENTIONS:
Other: Time restricted eating — 3 months (12 weeks) strict TRE intervention: Participants will be instructed to reduce their eating window by minimum 3 hours compared to habitual eating, with an eating window below 10 hours. The timing of the eating window is self-selected but should be placed between 6 am and 8 pm. Diet during the eating window is ad libitum with no further dietary restrictions.
  9 months (40 weeks) individually adjusted TRE intervention: An individual plan will be made based on participants' experiences during the strict TRE. Different choices of individual adjustment and support will be provided, including 1) eating window adjustments and the possibility of 'days off', 2) provision of a list of allowed calorie and caffeine free beverages that can be consumed outside the window, 3) continued opportunity to participate in peer-support group meetings, 4) extra phone calls with a project worker to discuss challenges or strategies to continue with TRE etc., and 5) further involvement of relatives.
  Arms: Time-restricted eating

SUMMARY:
The overall aim of the present study is to investigate the effectiveness of implementing a 1-year time-restricted eating (TRE)-based intervention on glycaemic control, body weight and composition, cardiometabolic risk factors, and behaviour in individuals with overweight/obesity and type 2 diabetes (T2D).

DETAILED DESCRIPTION:
In people with type 2 diabetes (T2D), weight loss is associated with improved glycaemic control and markers of cardiometabolic function as well as reduced use of antidiabetic medicine. Beyond pharmacological treatments, current strategies to reduce body weight and improve glycaemia include energy-restricted diets and increased physical activity.

Lifestyle interventions are complex, affecting many aspects of peoples' daily life. Dietary restrictions often result in rapid weight loss but the weight is gradually regained by many. Barriers to implement and maintain dietary changes include relapse of old habits and lack of knowledge, support, and insights into the type and amount of foods eaten. Previous lifestyle interventions targeting weight loss in T2D show efficacy for improving markers of metabolic and cardiovascular risk, including body weight and glycaemia during the intervention, but weight regain is often present. One reason may be that the intervention is not modified according to the needs of the target group. Often, weight loss interventions are shaped by a 'one size fits all' approach where both individual capabilities and motivation as well as social and contextual factors are more or less ignored. A user-based design could facilitate enrolment of participants and promote implementation and maintenance of the intervention among participants.

Intermittent fasting regimens have been suggested as efficient strategies for improving cardiometabolic health to a greater extent than can be attributed to the reduction in energy intake alone. TRE limits the time available for food intake to typically 8-10 hours/day without other dietary restrictions and has been put forward as a novel, acceptable, and safe strategy that has shown promising effects on body weight, glucose metabolism, appetite, and cardiometabolic health in individuals at high risk of T2D.

Although it has been suggested that TRE is a safe and feasible intervention, the longer-term effectiveness of TRE on glycaemic control and weight loss in individuals with T2D is unknown alongside the long-term acceptability and sustainability. Additionally, potential social and contextual challenges associated with integration of TRE into ordinary daily life structure and routines call for new approaches to support the individual in implementing and maintaining the strategy.

Overall, the RESET2 study consists of three phases; 1) Need assessment, 2) Pilot study, and 3) RCT. The aim of the present study (RCT) is to investigate the effectiveness of implementing a 1-year TRE-based intervention in individuals with overweight/obesity and T2D. Participants will attend 6 visits at Steno Diabetes Center Copenhagen (SDCC): Visit 0 (screening), Visit 1 (baseline, minimum 10 days after screening), Visit 2 (10 days prior to visit 3), Visit 3 [3 months (12 weeks) after baseline], Visit 4 (10 days prior to visit 5), Visit 5 [12 months (52 weeks) after baseline].

The specific objectives are:

1. To investigate the effect of a 1-year TRE intervention on changes in glycaemic control (HbA1c) in individuals with overweight/obesity and T2D.
2. To investigate the effects of a 1-year TRE intervention on changes in body weight, fat mass, continuous glucose monitoring (CGM) recorded time in range (TIR 3.9-10.0 mmol/l), and use of antidiabetic medication in individuals with overweight/obesity and T2D.
3. To describe changes in cardiometabolic risk factors (including fat-free mass, blood lipids, markers of kidney and liver function and inflammation, hormones involved in glucose metabolism and appetite control, liver fat, blood pressure, waist- and hip circumference), time below range (TBR), time above range (TAB), cognition, food preferences and reward, dim light melatonin onset (DLMO), and patient-reported outcomes including self-rated health, physical activity, well-being, diabetes distress, depression, food intake, and sleep quality.
4. To investigate the effects of a 3-month TRE intervention on changes in brain insulin sensitivity (sub-study).
5. To describe the extent to which the intervention was conducted as planned (visits, conversations, phone calls, peer support activities).
6. To describe the extent to which participants participated in support-related activities.
7. To explore participants' experiences with following TRE throughout a year including how they managed to keep their eating window and how the supporting activities and individualized approach worked for them (sub-population).
8. To explore the results from objectives 1-7 in relation to the extent the participants adhered to eating windows.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years
* Overweight or obesity (BMI ≥25 kg/m2)
* T2D with HbA1c>53 mmol/mol
* Habitual eating window ≥12 h/day (incl. foods/snacks and energy-containing beverages)

Exclusion Criteria:

* Bariatric surgery or planned bariatric surgery within study duration
* Use of fast acting insulin and combination insulin products
* Habitual CGM use
* A wish to adhere to Ramadan
* For women: current/planned pregnancy or lactation
* Alcohol or drug abuse (judged by investigator) or treatment with disulfiram
* Severe hypoglycaemia within last year (Severe hypoglycaemia, as defined by the American Diabetes Association (ADA), denotes severe cognitive impairment requiring external assistance for recovery)
* Inability to understand written and oral information in Danish
* Unable or unwilling to adhere to TRE; for instance, due to competing medical conditions.
* Medical condition which, based on investigators assessment, challenges participation including but not limited to severe heart, vascular or lung disease, cancer, chemotherapy, psychiatric, gastrointestinal, rheumatic, or endocrine diseases etc.
* Concomitant participation in other intervention study
* Inability to perform neuropsychological tests (e.g., severe vision and hearing impairment that can-not be improved with aids such as glasses and hearing aids, or language barrier.)

Exclusion criteria for the sub-study:

* Magnetic resonance imaging (MRI) contraindications based on the MR department's exclusion criteria including pacemaker or other implanted electronic devices, implanted metal objects not compatible to MRI scanning and severe claustrophobia
* Participants who do not wish to be informed about accidental findings by MR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c (mmol/mol) | Change from baseline to 3-months of intervention (strict TRE)
  Assessed from blood samples in fasted state.
Change in HbA1c (mmol/mol) | Change from baseline to the end of the intervention (12 months)
  Assessed from blood samples in fasted state.

SECONDARY OUTCOMES:
Body weight (kg) | Change from baseline to end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured on a digital scale in a fasted state.
Fat mass (kg) | Change from baseline to end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured by Dual-energy X-ray Absorptiometry in a fasted state.
Time in range (% 3.9-10.0 mmol/l) | Change from baseline to end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured using continous glucose monitoring.
Use of antidiabetic medication | Change from baseline to end of the intervention (12 months). Assessed at baseline, 3 months, 12 months.
  Change in current use of antidiabetic medication from baseline to end of the intervention (12 months).

OTHER OUTCOMES:
Body weight (kg) | Change from baseline to 3 months
  Measured on a digital scale in a fasted state.
Height (m) | Measured only at screening
  Height will be measured in order to calculate BMI.
Body mass index (kg/m^2) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Weight and height measurements will be used to calculate BMI in kg/m^2.
Fat mass (kg) | Change from baseline to 3 months
  Measured by Dual-energy X-ray Absorptiometry in a fasted state.
Time in range (% 3.9-10.0 mmol/l) | Change from baseline to 3 months
  Measured using continous glucose monitoring.
Use of antidiabetic medication | Change from baseline to 3 months
  Change in current use of antidiabetic medication from baseline to 3 months
Change in overall medication use | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Change in medication use (e.g. blood pressure, lipid-lowering medication etc)
Blood lipids (mmol/l) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentrations of: Total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides
Fat free mass (kg) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured by Dual-energy X-ray Absorptiometry in a fasted state.
Hormones-Insulin (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of insulin
Hormones-Glucagon (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of glucagon
Hormones-C-peptide (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of C-peptide
Hormones-Leptin (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of leptin
Hormones-Fibroblast growth factor 21 (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of fibroblast growth factor 21
Hormones-Glucagon-like peptide-1 (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of glucagon-like peptide-1
Hormones-Glucose-dependent insulinotropic polypeptide (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of glucose-dependent insulinotropic polypeptide
Hormones-Ghrelin (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of ghrelin
Hormones-Peptide YY (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of peptide YY
Hormones-Neuropeptide Y (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of neuropeptide Y
Hormones-Growth differentiating factor 15 (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of growth differentiating factor 15
Marker of kidney function - Creatinine (µmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of creatinine
Marker of kidney function - eGFR (mL/min) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Estimated glomerular filtration rate (eGFR)
Plasma beta-hydroxybutyrate (mmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of plasma beta-hydroxybutyrate
Marker of liver function - Aspartate-aminotransferase (U/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of aspartate-aminotransferase
Marker of liver function - Alanine aminotransferase (U/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of alanine-aminotransferase
Marker of liver function - Thrombocytes (x10^9/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of thrombocytes (for estimating liver-fibrosis)
Markers of inflammation- Tumor necrosis factor alpha (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of Tumor necrosis factor alpha
Markers of inflammation-Adiponectin (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of adiponectin
Markers of inflammation-C-reactive protein (mg/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of C-reactive protein
Markers of inflammation-Interleukin 6 (pmol/L) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Fasting concentration of interleukin 6
Time Below Range (% <3.9 mmol/l) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured using continous glucose monitoring.
Time Above Range (% >10.0 mmol/l) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured using continous glucose monitoring.
Coefficient of variation (CV) of glucose concentrations | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured using continous glucose monitoring.
Mean glucose concentrations | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured using continous glucose monitoring.
Standard deviation of glucose concentrations | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured using continous glucose monitoring.
Systolic blood pressure (mmHg) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured in a fasted and rest state.
Diastolic blood pressure (mmHg) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured in a fasted and rest state.
Resting heart rate (bpm) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured in a fasted and rest state.
Waist circumference (cm) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured using tape measure in a fasted state. The average of three consecutive measurements is reported.
Hip circumference (cm) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured using tape measure in a fasted state.The average of three consecutive measurements is reported.
Waist/hip ratio | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  The ratio of the circumference of the waist to that of the hips.
Degree of liver fibrosis (kPa) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured by FibroScan in a fasted state.
Degree of liver steatosis (dB/m) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured by FibroScan in a fasted state.
Food choice | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Food choice of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the Steno Biometric Food Preference Task (SBFPT). Food choice is determined based on frequency of selection made within each food category. The scores range from 0-48 i.e. 0 = foods within a specific food category have not been selected at all to 48 = foods within a specific food category have been selected 48 times.
Attention | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Measured using eye tracking in response to looking at food pictures during the SBFPT.
  Includes the following parameters: Gaze: Time spent (ms and %) and revisits (n); and fixations: Time to first fixation (ms), time spent (ms and %), fixation count (n), first fixation duration (ms), average fixation duration (ms). Distance to screen (mm), and gaze direction bias (ratio) which is calculated as the number of trials in which the first fixation was directed to a food image as a proportion to all trials. A bias score >0.5 indicates attention towards one food image, a bias score equal to 0.5 indicates no bias, and a bias score <0.5 indicates attention towards the other food images.
Reaction time (ms) | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Reaction time during forced food choice of food items from four combined food categories (high-fat savoury, high fat sweet, low-fat savoury and low-fat sweet foods) examined from the SBFPT.
Explicit liking | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Explicit liking of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the SBFPT. Explicit liking is rated using visual analogue scales (VAS) and the range is 0-100. Each end represents the extremes e.g. Question: "how pleasant would it be to taste this food right now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Explicit wanting | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Explicit wanting of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the SBFPT. Explicit wanting is rated using VAS and the range is 0-100. Each end represents the extremes e.g. Question: "how much do you want some of this food now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Implicit wanting | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Implicit wanting of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the SBFPT. Implicit wanting is assessed based on food choice and response time for selected and non-selected food items as well as mean response time (a frequency-weighted algorithm).
  In this frequency-weighted algorithm a positive score indicates a more rapid preference for a food type over another food type and a negative score indicates the opposite. A score of zero indicates that food types are equally preferred.The frequency weighted algorithm is used so the implicit wanting score is influenced by both selection (positively contributing to the score) and non-selection (negatively contributing to the score) of food type. Scores for implicit wanting typically range from -100-100 (due to reaction time there is no fixed min-max value).
Self-reported binge eating disorder | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Assessed from 2 questions (question 13,14) of Binge Eating Disorder Examination Questionnaire (EDE-Q 6.0).
Self-reported physical activity | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Assessed from the Physical Activity Scale 1 (PAS1)
Self-reported sleep quality | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Assessed from the Pittsburgh Sleep Quality Index (PSQI).The questionnaire consists of 19 items. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Self-reported information on social relations and social support | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Assessed from 2 items (items 68 and 70) of social relations and social support questionnaire (the Danish National Health Survey, item 68 and 70). The questions refer to contact with other people.
Self-reported sleepiness | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Assessed from the Epworth Sleepiness Scale (ESS).The questionnaire consists of 8 questions, which is weighted on a 0-3 interval scale. A low total score can be interpreted as a normal daytime sleepiness, and a higher score as a mild, moderate and severe excessive daytime sleepiness, respectively.
Self-reported eating behavior | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Assessed from the Dutch Eating Behavior Questionnaire (DEBQ). The questionnaire consists of 33 items and comprises three scales that measure emotional, external and restrained eating.Items can be rated from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behavior.
Self-reported night eating | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Assessed from the Night Eating Questionnaire (NEQ). The questionnaire consists of 14 items, that can be rated from 0 to 4. All items except item 13 are summed to obtain a global score. A total score ≥ 25 has been proposed as a lenient threshold for night eating syndrome.
Self-reported food intake | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Assessed from the food intake questionnaire (23-item FFQ). The questionnaire collects dietary data and uses a context-specific food list to estimate the usual diet.
Self-reported diabetes distress | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Assessed from the Problem Areas in Diabetes Scale (PAID-5 scale) comprising five of the emotional-distress questions of the full PAID items. Each item can be rated from 0 to 4. A total score of ≥ 8 indicates possible diabetes related emotional distress.
Self-reported sexual functioning/well-being | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Assessed from 1 item of the questionnaire the Danish National Health Survey (item 79) and 4 items of the questionnaire Danish PRO scheme (diabetes) (item 46 and 63-65).
Self-reported mood | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Assessed from the Major Depression Inventory (MDI). The questionnaire consists of 10 items. Each item can be rated from 0 to 5.The total score ranges from 0 to 50. A total score <20 indicates depression does not exist or its existence is doubtful, 20-24 indicates mild depression, 25-29 indicates moderate depression, and >29 indicates severe depression.
Self-assessed questionnaire to determine morningness-eveningness in human circadian rhythm | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Assessed by the Morningness-Eveningness Questionnaire (MEQ). The questionnaire consists of 19 items. Each item can be rated from 0 to 4-7. The total score ranges from 16 to 86. The lower score the more eveningness, and the higher score the more morningness.
Subjective appetite | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Subjective appetite will be assessed using Visual analogue scales (VAS), including ratings of hunger, fullness, satiety and prospective food consumption, thirst, desire to eat something sweet, salty, fatty, meat, and potential nausea.
Cognition | Change from baseline to 3 months and from baseline to the end of the intervention (12 months). Measured at baseline, 3 months, 12 months
  Cognitive functions will be assessed by Screen for Cognitive Impairment in Psychiatry Danish Version (SCIP-D) together with the Trail Making Test-Part B (psychomotor speed and executive function) and the Cognitive Failures Questionnaire
Dim light melatonin onset (DLMO) (subgroup only) | Change from baseline to 3 months. Measured at baseline and 3 months
  DLMO is a standard biomarker for measuring circadian rhythms and can easily be measured at home by saliva sampling. Saliva samples must be taken every 60 minutes under dim light (<30 lux) for at least 1 hour prior to and throughout the expected rise in melatonin.
Brain insulin resistance (subgroup only) | Change from baseline to 3 months. Assessed at baseline and 3 months.
  Cerebral blood flow assessed by MRI in response to intranasal insulin administration in a subgroup of participants. A basal MRI will be conducted and afterwards 160 U insulin will be administered intranasally by spraying 2 puffs per nostril (each containing 10 U of insulin) every minute over 4 minutes followed by MRI 30 minutes after the last administration
Adherence (%) | Registered 2 days/week on random days via an online questionnaire.
  Degree of adherence to eating windows = (number of days where eating window was reduced by minimum 3 hours compared to habitual eating window and participants have reported an eating window below 10 hours / total number of days in intervention) * 100%.
Degree of participants' participation in intervention activities - Visits | Visit 1, visit 2, visit 3, visit 4, visit 5
  Assessed from % participation in the 5 intervention visits
Degree of participants' participation in intervention activities - Conversations | Conversations at visit 1 and visit 3
  Assessed from % participation in the conversations at visit 1 and 3 (TRE group only)
Degree of participants' participation in intervention activities - Peer support group meetings | Support group meetings will be held once monthly
  Assessed from % participation in peer support group meetings (TRE group only)
Degree of participants' participation in intervention activities - Phone calls | Phone calls after 2, 6, 9 weeks + Phone calls after 6 and 9 months
  Assessed from % participation in the phone calls (TRE group only)
Participants' acceptance of TRE | The interviews will be conducted at the end of intervention (1 year after baseline) at visit 5
  Assessed by interviews on participants' acceptance of TRE in terms of bodily/physical experiences, motivation, and ability to manage TRE in daily living and how intervention activities were supportive. This refers only to the TRE group. Individual interviews will be conducted by a qualitative researcher with a sub-group of participants in the TRE group (n=30) representing experiences with a variety of individual adjustments after the last visit, and focus group interviews will be performed with a sub-group of participants in the TRE group (n=30) choosing peer support or family involvement. Participants are free to say yes or no to participate in interviews.These interviews will be audio recorded.
Energy intake (kJ) | Registrations prior to baseline (visit 1), after 3 months (visit 3), and after 12 months (visit 5)
  Assessed from 3-day dietary records
Fat energy percent | Registrations prior to baseline (visit 1), after 3 months (visit 3), and after 12 months (visit 5)
  Assessed from 3-day dietary records
Carbohydrate energy percent | Registrations prior to baseline (visit 1), after 3 months (visit 3), and after 12 months (visit 5)
  Assessed from 3-day dietary records
Protein energy percent | Registrations prior to baseline (visit 1), after 3 months (visit 3), and after 12 months (visit 5)
  Assessed from 3-day dietary records
Alcohol energy percent | Registrations prior to baseline (visit 1), after 3 months (visit 3), and after 12 months (visit 5)
  Assessed from 3-day dietary records
Dietary fibers (gram) | Registrations prior to baseline (visit 1), after 3 months (visit 3), and after 12 months (visit 5)
  Assessed from 3-day dietary records

CONTACTS AND LOCATIONS:
Overall Officials: Jonas S Quist, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No